CLINICAL TRIAL: NCT03230604
Title: Clinical Performance of Bulk-fill Resins Composite Restorations on Posterior Tooth of Adults Patients. Randomized Doble-blind Trial
Brief Title: Clinical Performance of Two Bulk-Fill Composite of Posterior Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Patricio Vildosola Grez, Associate Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DI-1301-16/CB
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Post Dental Restoration; Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Intervention: Bulk full composite (3M) bulk fill composite in posterior class one cavities bulk fill composite in posterior class two cavities bulk fill composite in posterior class five cavities
  Intervention:Bulk full composite (Ivoclar-Vivadent) bulk fill composite in posterior class one cavities bulk fill composite in posterior class two cavities bulk fill composite in posterior class five cavities Other: bulk fill composite Intervention Control: Nano resin composite (K Z350 xt) Restoration in class one cavities Restoration in class Two cavities Restoration in class five cavities
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulk-Fill composite Class I, II and V cavities (Active Comparator): Restorative with Filtek Bulkfill composite in class I, II and V Restorative with Tetric N Ceram composite in class I, II and V
  Interventions: Device: Filtek Bulk Fill Composite and Tetric N Ceram Bulk Fill Composite; Device: Z 350 Xt Composite
- Z 350 xt Composite (Active Comparator): Restorative with Z 350 xt composite in class I, II and V
  Interventions: Device: Filtek Bulk Fill Composite and Tetric N Ceram Bulk Fill Composite; Device: Z 350 Xt Composite

INTERVENTIONS:
Device: Filtek Bulk Fill Composite and Tetric N Ceram Bulk Fill Composite — Restorative cavities one, two and five with material Filtek Bulk Fill Composite
Device: Z 350 Xt Composite — Restorative cavities one, two and five with material Z 350 XT Composite

SUMMARY:
To minimize the effects of polymerization shrinkage in the restorative treatment, there are new composites called Bulk- Fill which the companies has developed this composites for example Tetric N Ceram(Ivoclar-Vivadent) and Filtek ( 3M ESPE). Its decreased polymerization shrinkage and properties allow the material to be inserted in one layer being quickly than traditional composite. This clinical study is designed to compare the clinical performance of the bulk fill composite resin in Class I (one-surface posterior), II (two-surface posterior) and V (cervical-surface posterior) fillings.

DETAILED DESCRIPTION:
A patients with 3 caries lesions class one either two or five will be divided into 3 groups , cavities will be incrementally layered with resin composite and each increment will be cured as directed by the manufacturer with the light curing unit (Bluephase Style Ivoclar-Vivadent), with an energy 1,100 mW/cm² (±50 mw/cm²) and others group of cavities will be restored by bulk fill composite (3M ESPE) and other bulk fill composite ( IVOCLAR-VIVADENT) as one increment then will be cured as directed by the manufacturer with the light curing unit.

The study will investigate the clinical performance and efficacy of a bulk-filled composite resin restorative material for a period of 5 years

ELIGIBILITY:
Inclusion Criteria:

* must have given written informed consent to participate in the trial
* need at least three posterior restorations
* must be available for the required post-operative follow-up visits
* have a buccal to lingual/palatal width no greater than 1/3 the distance from buccal to lingual/palatal cusp tips
* At least one occlusal and proximal contact on a natural tooth
* Cavities depth > 2 mm in cervico-occlusal

Exclusion Criteria:

* have severe medical complications (organ transplants, long term antibiotic or steroid treatment, cancer or immunocompromised) and disabilities who may not be able to tolerate the time required to complete the restorations
* have xerostomia either by taking medications known to produce xerostomia or those with radiation induced or Sjogren's syndrome patients
* chronic periodontitis
* present with any systemic or local disorders that contra-indicate the dental procedures included in this study
* an unstable occlusion
* severe bruxing
* teeth with periapical pathology or expected pulp exposures
* are pregnant.
* Endodontically treated teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance restoration | six month, one years, two, three, four and five years
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI criteria , Unit is Ranking system has 5 scores for each different criterion. Either restoration is clinically excellent, or good, or sufficient, or unsatisfactory, or clinically poor.

CONTACTS AND LOCATIONS:
Overall Officials: Odontologia, Principal Investigator — Universidad Andres Bello
Locations (1):
- Patricio Vildosola Grez, Santiago, Santiago Metropolitan, Chile